CLINICAL TRIAL: NCT03451318
Title: A Multicenter Study of Establishing the Multi-disciplinary Cooperative Diagnosis and Treatment Process and Evaluation System for Children With Sleep Disordered Breathing and Malocclusion
Brief Title: Multi-disciplinary Diagnosis and Treatment Process and Evaluation System for Children With Sleep Disordered Breathing and Malocclusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Stomotological Hospital (Other)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Shanghai Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16CR2044B
Record Dates: First submitted 2018-02-07; First posted 2018-03-01 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) and Malocclusion
MeSH Terms: conditions — Sleep Apnea, Obstructive; Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- drug therapy (Active Comparator): Nasonex(mometasone furoate),1 spray,QD (Quaque Die in Latin),for 3 months.
  Interventions: Drug: Mometasone Furoate Nasal Spray
- tonsillar adenoidectomy (Active Comparator): tonsillar adenoidectomy
  Interventions: Procedure: tonsillar adenoidectomy
- orthodontic treatment (Active Comparator): Apply Twin-block appliance combined with maxillary expander
  Interventions: Procedure: Maxillary expander plus Twin-Block
- tonsillar adenoidectomy plus orthodontic treatment (Active Comparator): Apply Twin-block appliance combined with maxillary expander one month after tonsillar adenoidectomy .
  Interventions: Procedure: tonsillar adenoidectomy; Procedure: Maxillary expander plus Twin-Block

INTERVENTIONS:
Drug: Mometasone Furoate Nasal Spray — Mometasone Furoate Nasal Spray NASONEX
  Arms: drug therapy
Procedure: tonsillar adenoidectomy — tonsillar adenoidectomy
  Arms: tonsillar adenoidectomy; tonsillar adenoidectomy plus orthodontic treatment
Procedure: Maxillary expander plus Twin-Block — Twin-block appliance combined with maxillary expander
  Arms: orthodontic treatment; tonsillar adenoidectomy plus orthodontic treatment

SUMMARY:
The aim of this study is to compare the efficacy and safety of drug therapy, tonsillar adenoidectomy only, orthodontic treatment only and tonsillar adenoidectomy plus orthodontic treatment in children with obstructive sleep apnea hypopnea syndrome (OSAHS) and malocclusion.

In this study, we hope to improve children's OSAH in function, three-dimensional shape and subjective and objective symptoms of sleep breathing through tonsillar adenoidectomy plus orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as mild to moderate OSAHS
2. Tonsil and/or adenoid hypertrophy
3. Narrow dental arch and / or mandibular retrusion (ANB value≥ 4.5)
4. The guardian / child can understand the study and sign the informed consent

Exclusion Criteria:

1. Patients with nasal obstruction disease
2. The pathological obesity
3. Patients with systemic disease
4. Patient with central sleep apnea/hypopnea syndrome

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2018-03-02 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Obstructive Apnea Index（OAI）/ Apnea Hypopnea Index （AHI） in PolySomnoGraphy （PSG） | change from baseline at 7 months,1 year & 2 years post-treatment
  OAI/AHI (which are in negative correlation with oxygen saturation) decrease after treatment

SECONDARY OUTCOMES:
Low arterial Oxygen Saturation （LSaO2） in PSG | change from baseline at 7 months,1 year & 2 years post-treatment
  LSaO2 increase after treatment
Airway volume change as shown on Cone Beam Computer Tomography (CBCT) | change from baseline at 7 months post-treatment
  Airway volume increase after treatment
ANB, Frankfort plane- Mandibular plane Angle (FMA) measurement using X-ray cephalometrics. | change from baseline at 7 months,1 year & 2 years post-treatment
  ANB & FMA (face development indicators) become normal after treatment
Assessment of subjective efficacy by using a "questionnaire on children's sleep symptoms" | change from baseline at 7 months,1 year & 2 years post-treatment
  Sleep quality improve after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yuehua Liu, Professor, Principal Investigator — Department of Orthodonitcs,Shanghai Stomatological Hospital
Locations (1):
- Shanghai Stomotological Hospital, Shanghai, China

REFERENCES:
- [Derived] Li Y, Wu J, Guo J, Yu L, Wang J, Li X, Xu S, Zhu M, Feng J, Liu Y. The efficacy of different treatment approaches for pediatric OSAHS patients with mandibular retrognathia: study protocol for a multicenter randomized controlled trial. Trials. 2020 Jun 30;21(1):595. doi: 10.1186/s13063-020-04398-9. PMID 32605655